CLINICAL TRIAL: NCT05807165
Title: Hypofractionated Stereotactic Radiotherapy Versus Hippocampus-sparing Whole-brain Radiotherapy in Treating Cancer Patients With Brain Oligometastases: A Phase II Parallel Non-randomized and Prospective Observational Study
Brief Title: HF-SRT vs. HS-WBRT in Treating Patients With Brain Oligometastases
Status: Not yet recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202201915A3
Record Dates: First submitted 2023-03-05; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-12

CONDITIONS: Brain Oligometastases
Keywords: Brain Oligometastases; Stereotactic Radiotherapy (SRT); Hypofractionation; Hypofractionated Stereotactic Radiotherapy (HF-SRT); Hippocampus; Hippocampus-Sparing Whole-Brain Radiotherapy (HS-WBRT); Neurocognitive Functions (NCFs); Central Nervous System (CNS); Progression-free Survival (PFS); CNS Progression-Free Survival (CNS-PFS); Patterns of CNS Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HF-SRT: RT techniques and the dose schemes in the cohort of Hypofractionated Stereotactic Radiotherapy (HF-SRT)
  Interventions: Radiation: Hypofractionated Stereotactic Radiotherapy (HF-SRT)
- HS-WBRT plus memantine: The course of hippocampus-sparing whole-brain radiotherapy (HS-WBRT) combined with the synergic use of the neuroprotective agent, memantine
  Interventions: Radiation: Hippocampus-Sparing Whole-Brain Radiotherapy (HS-WBRT) plus memantine

INTERVENTIONS:
Radiation: Hypofractionated Stereotactic Radiotherapy (HF-SRT) — The administered dose-fractionation schemes range between 30 and 35 Gy delivered within two weeks with a dose per fractionation ranging from 6 to 7 Gy.
  Groups: HF-SRT
Radiation: Hippocampus-Sparing Whole-Brain Radiotherapy (HS-WBRT) plus memantine — * The prescribed dose is 30 Gy delivered in 12 fractions for therapeutic or adjuvant WBRT.
  * The prescription of memantine for finally twice-daily dosing will be prescribed as follows:
    * During the first 3 weeks concurrent with the delivery of hippocampus-sparing WBRT, 5-mg morning dose will be initially prescribed [Week 1 -3]
    * 5-mg twice a day in the following week [Week 4]
    * A morning dose of 10 mg and an evening dose of 5 mg in the following week [Week 5]
    * 10-mg twice a day for the subsequent weeks up to Week 24 [Week 6 - 24]
  Groups: HS-WBRT plus memantine

SUMMARY:
[Background] For newly-diagnosed patients with brain metastases (BMs), conventional whole-brain radiotherapy (WBRT) might still remain a common palliative management. However, WBRT-related late consequences, particularly a decline in neurocognitive functions (NCFs), are a major concern. Actually, WBRT-related neurocognitive dysfunction is usually characterized as deterioration involving learning and memory, in which the extremely radiosensitive hippocampus indeed plays a critical role.

To postpone the occurrence and mitigate neurocognitive impairments associated with conventional WBRT, there have been some strategies in the clinical practice of radiation oncology. Among them, the technology/technique of highly precise/accurate stereotactic radiosurgery or stereotactic radiotherapy (i.e., hypofractionated stereotactic radiotherapy, HS-SRT) might have been widely administered in irradiating exclusively the focal brain metastatic lesions, particularly in cancer patients with a limited number of brain metastases. By contrast, the planning strategy of hippocampus avoidance during the course of whole-brain irradiation has also been well-established in preserving NCFs.

[Methods] Newly-diagnosed cancer patients harboring 1 - 4 brain metastatic lesions are eligible if they still have fair/good performance status. Eligible and enrolled should receive baseline brain MRI examination and pre-WBRT neurocognitive assessment. Although non-randomized, this phase II trial comprises two prospective (radiotherapeutic) cohorts with individually different planning techniques and prescription schedules. Cohort I represents patients referred for arranging partial-brain irradiation; namely, a course of hypofractionated stereotactic radiotherapy (HF-SRT) is delivered within 2 weeks with a cumulative dose of 3000 - 3500 cGy in 5 fractions. By contrast, Cohort II stands for patients referred for arranging the course of hippocampus-sparing WBRT (HS-WBRT), delivered within 3 weeks with a cumulative dose of 3000 cGy in 12 fractions, during which the planning technique of simultaneous integrated boost (SIB) is employed to focally escalate the dose irradiating the brain metastatic foci. Besides, adhering to several international clinical practice guidelines, the synergic use of the neuroprotective agent (memantine) will be routinely applied in the treatment Cohort II (HS-WBRT). In both treatment cohorts, a battery of neuropsychological measures, which includes 7 standardized neuropsychological tests (e.g., executive functions, verbal and non-verbal memory, working memory, and psychomotor speed), is used to evaluate neurocognitive functions.

The primary outcome measure is the median time of CNS progression-free survival (CNS-PFS). Secondary outcome measures encompass both neuro-oncological endpoints and neurocognitive endpoints, among which there is cognitive-deterioration-free survival (CD-free survival). CD-free survival is defined mainly as the time from enrollment to a NCF decline of exceeding than 1 SD away from the baseline involving at least one of the assessed NCF tests. Additionally, patients who expire before 6 months or are alive but fail to undergo all the neurocognitive testing administered would also be defined as suffering from cognitive deterioration.

[Expected results] This prospective observational study aims to examine thoroughly and analyze the comparatively between the two radiotherapeutic cohorts (HF-SRT versus HS-WBRT), addressing both CNS tumor control and neurocognitive functional outcomes. It is expected that the patterns of (CNS) failure and individual time to progression will be clearly demonstrated in this prospective observational study encompassing two distinct radiotherapeutic cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically-confirmed non-hematopoietic malignancy who are referred for postoperative adjuvant or therapeutic hypofractionated stereotactic radiotherapy (HF-SRT)
* A Fair/good performance status no worse than Eastern Cooperative Group (ECOG) of 2 or an acceptable performance status of Karnofsky Score (KPS) at least 70
* The number and extent of brain metastatic lesions should be no more than three metastatic foci with a greatest diameter no more than 4 cm shown on pre-radiotherapy MRI; namely, that is the clinical setting of oligometastatic brain disease or brain oligometastases

Exclusion Criteria:

* Patients with their primary cancer arising from hematological malignancies (i.e., malignant lymphomas, leukemia), germ cell tumors, or malignant meningiomas
* Patients with MRI-identified metastasis within 5 mm peri-hippocampally
* Patients with metastasis involving the brain stem
* Clinical suspicion of leptomeningeal spreading
* History of prior radiotherapy including stereotactic radiosurgery delivered to brain/head region for any reasons

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with newly-diagnosed brain oligometastases and an acceptable performance status would receive baseline neurocognitive assessment.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
CNS progression-free survival (CNS-PFS) | The time from study enrollment to CNS disease progression of death from any cause, assessed up to 10 years.
  The median CNS progression-free survival (CNS-PFS), which is a time-dependent endpoint, defined as the time from study enrollment to CNS disease progression of death from any cause.
Cognitive-deterioration-free survival (CD-free survival) | The time from enrollment to a cognitive decline of exceeding more than 1SD away from the baseline in at least one of the assessed NCF tests, assessed up to 24 months.
  The time from enrollment to a cognitive decline of exceeding more than 1SD away from the baseline in at least one of the assessed NCF tests. Furthermore, regarding cognitive-deterioration-free survival, patients who expire before 6 months or are alive but do not undergo all the neurocognitive testing administered or even fail to receive MMSE evaluation would be assumed reasonably that they suffer cognitive deterioration at the time of death or at the time point, or they fail to receive their first neurocognitive assessment follow-up as long as there are no subsequent NCF assessments.

SECONDARY OUTCOMES:
Overall survival (OS) | The time from enrollment to death, assessed up to 10 years.
Median survival time (MST) | The time from enrollment to death, assessed up to 10 years.
Causes of death (neurologic vs non-neurologic death) | The time from enrollment to death, assessed up to 10 years.
Patterns of CNS (Intracranial or Leptomeningeal Disease) failure evaluated through brain MRI | The time from enrollment to CNS failure, assessed up to 10 years.
  Three patterns of central nervous system (CNS) failure were classified particularly when the CNS progression in the corresponding patient manifests for the first time after the course of HF-SRT: intracranial local failure (LF), distant brain parenchymal failure (DPF), and development of leptomeningeal disease (LMD).
Time to progression (TTP) | The time from enrollment to CNS progression, assessed up to 10 years.
  Time to CNS progression
Progression-free survival (PFS) | The time from enrollment to disease progression, assessed up to 10 years.
  Intracranial PFS or CNS progression-free survival; CNS progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan